CLINICAL TRIAL: NCT04179305
Title: Giving Information Systematically and Transparently in Lung and GI Cancer Phase 2
Acronym: Oncolo-GIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-07020392-Phase2; R21NR018693 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Critical Illness; Oncology; Communication
MeSH Terms: conditions — Critical Illness; Neoplasms; Communication

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oncolo-GIST Arm - Patients (Experimental): Patients assigned to this arm will discuss scan results revealing progressive disease with an Oncolo-GIST trained physician.
  Oncolo-GIST: Behavioral: Oncolo-GIST Oncolo-GIST is a brief, manualized communication intervention that guides oncologists in "gist communication" by itemizing 4 key steps in the process of imparting prognostic information.
  Topics covered include:
  Principles of introducing prognosis in the setting of worsened scan results Coupling communicating realistic prognoses with psychological support (e.g., saying "average life-expectancy is months…" with emphasizing that the oncology team "will always provide care for you") Addressing informational needs and psychological reactions Applying proven techniques for supporting patients who are reluctant to discuss prognosis.
  Interventions: Behavioral: Oncolo-GIST
- Usual Care Arm - Patients (Placebo Comparator): Patients assigned to this arm will will discuss scan results revealing progressive disease with a physician that was not trained with the Oncolo-GIST intervention.
  Usual Care Arm: Oncologists will provide care in non-specific manner.
  Interventions: Behavioral: Usual Care Arm
- Oncolo-GIST Arm - Physicians (Experimental): Physicians assigned to this arm will receive the Oncolo-GIST training intervention.
  Interventions: Behavioral: Oncolo-GIST
- Usual Care Arm - Physicians (Placebo Comparator): Physicians assigned to this arm will not receive the Oncolo-GIST training intervention.
  Interventions: Behavioral: Usual Care Arm

INTERVENTIONS:
Behavioral: Oncolo-GIST — Behavioral: Oncolo-GIST Oncolo-GIST is a brief, manualized communication intervention that guides oncologists in "gist communication" by itemizing 4 key steps in the process of imparting prognostic information.
  Topics covered include:
  Principles of introducing prognosis in the setting of worsened scan results Coupling communicating realistic prognoses with psychological support (e.g., saying "average life-expectancy is months…" with emphasizing that the oncology team "will always provide care for you") Addressing informational needs and psychological reactions Applying proven techniques for supporting patients who are reluctant to discuss prognosis.
  The 4-step guide will include brief video-clips of demonstrating each "talking point" with a standardized patient, including ideal scenarios, common pitfalls to avoid, and how to respond to patient reactions that are particularly challenging, such as responding to optimism, death anxiety, and reliance on faith.
  Arms: Oncolo-GIST Arm - Patients; Oncolo-GIST Arm - Physicians
Behavioral: Usual Care Arm — Oncologists will provide care in non-specific manner.
  Arms: Usual Care Arm - Patients; Usual Care Arm - Physicians

SUMMARY:
When advanced disease progresses, there comes a time when an oncologists must explain to their patients that they only have months left to live. During these discussions the oncologist attempts to explain to the patient their prognoses and what it means for them going forward. However our prior studies shown that even when patients only have months left to live, most do not understand that their cancer is incurable and that it is late/end-stage.

Dying cancer patients who fully understand their prognosis are able to make more informed decisions and are therefore more likely to engage in advanced care planning, and receive care what in consistent with their values and preferences. They are also in a better position to avoid burdensome, non-beneficial care. The investigator developed Oncolo-GIST in order to help increase the number of patients who fully understand their prognosis and its implications.

Oncolo-GIST is an intervention aimed at enhancing clinicians' communication with patients by teaching them to relay information both sensitively and using simple terminology. The Oncolo-GIST training will provide instruction in areas such as how to introduce the topic of prognosis (describe scan results as "worse"), how to phrase the prognosis itself ("likely months, not years"), how to explain expected treatment outcomes (e.g., "not expected to be cured by treatment") and how to describe expected treatments impact on quality of life - that is, whether the anticancer treatment is likely to make them feel overall better or worse. The training materials consist of a manual and a set of videos that act out situations described in the manual.

The second phase of this study will be a randomized controlled trial. The investigator will recruit (n=50) adults with metastatic GI or lung cancers with scan results that reveal progression (worsened disease) on an initial systemic treatment; that is, patients whose life-expectancy can reliably be estimated to be months, not years. Medical oncologists (n=4) who care for these patients will also be consented for study participation and half (n=2) will be randomized to receive the Oncolo-GIST training.

Patients will be assessed by trained research staff in the week prior to a scheduled meeting with their oncologist to discuss the scan results. This will provide patients' baseline levels of prognostic understanding and enable the investigator to determine how the intervention relates to pre-post scan visit changes in prognostic understanding. Patients will be assessed post-scan within a week of that progressive scan visit.

The assessment battery that will be administered at these time-points will measure the patient's degree of prognostic understanding, the primary outcome of the study. Other outcomes that will be measured by the assessment battery include the patients quality of life, therapeutic alliances of the patient, whether or not a DNR was ordered, the care received by the patient, whether or not the patient preferred greater quality of longer quantity of life, and whether or not the patients received "value-consistent" care.

DETAILED DESCRIPTION:
Despite exciting recent advances in cancer treatments, there still, ultimately, comes a time when advanced disease progresses, and patients can reliably be expected to have months, not years, left to live. For patients with metastatic cancers studied in the investigator's Coping with Cancer NCI R01s, this comes after progression on 1st- or 2nd-line therapy -- be it chemo-, immune-, or targeted therapy. Prior studies conducted by the investigator have found that oncologists can reliably predict when patients have only months to live (e.g., remarkable agreement between oncologist estimates of months to live shared with patients and patients' actual survival of months). By contrast, patients appear largely unaware of their prognosis. For example, 5% of patients a median of 5 months from death, accurately understood they had incurable, late/end-stage, terminal cancer, and likely only months to live. Dying cancer patients appear to lack the prognostic understanding needed to make informed choices.

Patients who grasp that they are dying (e.g., the 8.6% who "get the gist" that they likely have months to live), relative to those who do not, have been shown to have: a) higher rates of advance care planning (ACP), b) receive less burdensome, unbeneficial care (e.g., fewer intensive care unit, ICU, stays, less cardiopulmonary resuscitation, CPR), and c) more value-consistent care. The investigator has found that patient prognostic understanding is improved by oncologist discussions of life-expectancy, but despite 71% of patients wanting to discuss prognosis with their oncologists (83% adult cancer patients thought prognostic information was extremely/very important), only 17.6% of cancer patients within months of death reported that they had discussed prognosis with their oncologist. Not only do oncologists appear to discuss prognosis less than patients want them to, but even when prognostic discussions do occur, the investigator has found that some approaches (e.g., matter-of-fact) are more effective than others (e.g., vague) for promoting patients' prognostic understanding. Thus, prior work identifies a need to improve communication to promote patient prognostic understanding in a way that oncologists will likely learn, accept, use, and possibly implement more broadly in clinical practice.

To address this need, the investigator developed the "Giving Information Simply &Transparently" (GIST), Oncolo-GIST intervention -- a manualized oncologist communication intervention that simplifies how to impart prognostic information by focusing on 4 basic steps: 1) Giving scan information, 2) Informing prognosis, 3) Strategizing sensitively, and 4) Transparently asking what the patient heard. Unlike traditional emphasis on numerical or medical details, the Oncolo-GIST approach is based on Reyna's Fuzzy-Trace Theory of decision-making, which emphasizes the need for an understanding of the bottom-line gist of a situation. The Oncolo-GIST approach distills prognostic discussions to clear communication of end-of-life (EoL) decision-making essentials (e.g., life-expectancy). 3 specific aims of the Oncolo-GIST approach will be tested in 2 phases:

Phase 1 will consist of two parts: 1) An interview of key stakeholders/key informants regarding Oncolo-GIST Version 1.0 in order to inform refinements to produce Oncolo-GIST Version 2.0. 2) An open trial of Oncolo-GIST Version 1.0 to inform refinements to produce Oncolo-GIST Version 2.0.

Phase 2 will involve a cluster randomized controlled trial (RCT) of Oncolo-GIST Version 2.0 on 50 patients with metastatic cancers worse on at least 1 line of therapy (chemo-, immune-, targeted), whose oncologists do not expect them to survive 12 months. Patients will be assessed in the week prior to their scheduled scan, within 1 week of the clinic visit in which progressive scan results are discussed, and then 2 and 4 months later to explore intervention effects on primary and secondary outcomes, respectively. Oncologists will be assessed in the week following that same clinic visit to obtain their impressions of the discussion of prognosis and the patient's prognostic understanding.

In Phase 2, for the pilot cluster RCT, the investigator will recruit (n=50) adults with metastatic GI or lung cancers with scan results that reveal progression (worsened disease) on an initial systemic treatment; that is, patients whose life-expectancy can reliably be estimated to be months, as opposed to years. Medical oncologists (n=4) who care for these patients will also be consented for study participation and half (n=2) will be randomized to receive the Oncolo-GIST training. The investigator expects 12-13 patients will be clustered within each of the 4 oncologists. Hierarchical Linear Modeling (HLM) techniques will be employed to address the non-independence of patient assessments within each cluster. Patients (n=25) will be seen by either an Oncolo-GIST trained oncologist or an oncologist not trained in the intervention; that is, usual care (n=25). Patients in both arms will have met the same eligibility criteria (i.e., have similar prognoses).

Patients will be assessed by trained research staff in the week prior to a scheduled meeting with their oncologist to discuss the scan results. This will provide patients' baseline levels of prognostic understanding and enable the investigator to determine how the intervention relates to pre-post scan visit changes in prognostic understanding. Patients will be assessed post-scan within a week of that progressive scan visit. Although not all patients are expected to die within the study observation period, given a median life expectancy of ~4-5 months from baseline, the investigator expects nearly half of the enrolled patients will die 4 months from baseline, and that the vast majority will die during the study observation period of 12 months. Thus, for all patients enrolled in this study, the medical care that they receive can reasonably be considered end-of-life care, whether they die during the study observation period or not.

The primary outcome is the patient's degree of prognostic understanding, measured using the investigator's validated 4-item assessment. The investigator will determine if the patient understood the scan results to be "worse" and their understanding of expected outcomes of treatments proffered (re: curability, survival, quality of life). Outcomes will also include whether a DNR order was completed for the patient, the McGill Quality of Life measure, performance status (e.g., Eastern Cooperative Oncology Group, ECOG), and care received (e.g., anticancer, intensive, palliative care). Treatment preferences will be assessed using the SUPPORT question regarding quality vs. quantity of life, which will be used to compare with actual EoL care received to operationalize "value-consistent" care. The investigator's validated Human Connection scale will assess therapeutic alliances from both the patient and oncologist perspective, and the investigator will assess oncologists' sense of how the scan discussion went (e.g., degree to which they think they communicated effectively, and that the patient understood them and had an accurate prognostic understanding). Demographic/background information (e.g., age, race/ethnicity, sex, education) and DNR documentation will be obtained from subject self-report at baseline and the patient's medical records. Previously validated measures will assess potential confounding influences such as time from diagnosis, prior discussions of prognosis, and health literacy using the REALM. Preferences regarding medical decision-making (e.g., an active vs. passive role in deciding the best course of treatment), patients' Religious Beliefs in EoL Care (RBEC), and the question "If your doctor knew how long you had left to live, would you want him/her to tell you?" will be assessed.

Hierarchical Linear Modeling (HLM) will be used to evaluate intervention effects. HLM is statistically appropriate because it accounts for the clustering of patients within oncologists, creating non- independence of clustered assessments. HLM will model oncologists as a random effect as has been done in prior RCTs. Baseline covariates known to affect study outcomes (e.g., patient health literacy) will be included in models to increase the precision of effect size estimates. This will provide a preliminary effect size estimate of Oncolo-GIST Version 2.0's ability to improve patients' prognostic understanding for a future, larger study. Linear and logistic regression models will estimate effects of the Oncolo-GIST intervention on secondary and exploratory outcomes.

The details for Phase 1 of the study are enumerated in a separate record marked "Giving Information Systematically and Transparently in Lung and GI Cancer Phase 1" (Oncolo-GIST P1) with NCT # NCT04158908.

ELIGIBILITY:
Clinicians

Inclusion Criteria:

* Specialize in Lung and GI cancers
* Currently provide care at the WCM Lung and GI cancer clinics
* Fluent in English

Exclusion Criteria:

* Does not specialize in Lung and GI cancers
* Does not currently provide care at the WCM Lung and GI cancer clinics
* Not fluent in English

Patients

Inclusion Criteria:

* Receiving ongoing care (≥ 2 visits) that includes regular scans
* Progression on at least 1 line of systemic cancer therapy
* Prognosis from an oncologist of less than 12 months
* Receiving care from an oncologist participating in the Oncolo-GIST study
* Fluent in English

Exclusion Criteria:

* Does not specialize in Lung and GI cancers
* Does not currently provide care at the WCM Lung and GI cancer clinics
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly G Prigerson, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambden J, Zhang B, Friedlander R, Prigerson HG. Accuracy of Oncologists' Life-Expectancy Estimates Recalled by Their Advanced Cancer Patients: Correlates and Outcomes. J Palliat Med. 2016 Dec;19(12):1296-1303. doi: 10.1089/jpm.2016.0121. Epub 2016 Aug 30. PMID 27574869
- [Background] Enzinger AC, Zhang B, Schrag D, Prigerson HG. Outcomes of Prognostic Disclosure: Associations With Prognostic Understanding, Distress, and Relationship With Physician Among Patients With Advanced Cancer. J Clin Oncol. 2015 Nov 10;33(32):3809-16. doi: 10.1200/JCO.2015.61.9239. Epub 2015 Oct 5. PMID 26438121
- [Background] Epstein AS, Prigerson HG, O'Reilly EM, Maciejewski PK. Discussions of Life Expectancy and Changes in Illness Understanding in Patients With Advanced Cancer. J Clin Oncol. 2016 Jul 10;34(20):2398-403. doi: 10.1200/JCO.2015.63.6696. Epub 2016 May 23. PMID 27217454
- [Background] Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. J Clin Oncol. 2010 Mar 1;28(7):1203-8. doi: 10.1200/JCO.2009.25.4672. Epub 2010 Feb 1. PMID 20124172
- [Background] Wright AA, Zhang B, Keating NL, Weeks JC, Prigerson HG. Associations between palliative chemotherapy and adult cancer patients' end of life care and place of death: prospective cohort study. BMJ. 2014 Mar 4;348:g1219. doi: 10.1136/bmj.g1219. PMID 24594868
- [Background] Prigerson HG. Socialization to dying: social determinants of death acknowledgement and treatment among terminally ill geriatric patients. J Health Soc Behav. 1992 Dec;33(4):378-95. PMID 1464721
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Mack JW, Fasciano KM, Block SD. Communication About Prognosis With Adolescent and Young Adult Patients With Cancer: Information Needs, Prognostic Awareness, and Outcomes of Disclosure. J Clin Oncol. 2018 Jun 20;36(18):1861-1867. doi: 10.1200/JCO.2018.78.2128. Epub 2018 Apr 23. PMID 29683788
- [Background] Reyna VF. Theories of medical decision making and health: an evidence-based approach. Med Decis Making. 2008 Nov-Dec;28(6):829-33. doi: 10.1177/0272989X08327069. No abstract available. PMID 19020341
- [Background] Elsayyad A. Informed consent for comparative effectiveness trials. N Engl J Med. 2014 May 15;370(20):1958-9. doi: 10.1056/NEJMc1403310. No abstract available. PMID 24827054
- [Background] Spellecy R, Tarima S, Denzen E, Moore H, Abhyankar S, Dawson P, Foley A, Gersten I, Horwitz M, Idossa L, Joffe S, Kamani N, King R, Lazaryan A, Morris L, Horowitz MM, Majhail NS. Easy-to-Read Informed Consent Form for Hematopoietic Cell Transplantation Clinical Trials: Results from the Blood and Marrow Transplant Clinical Trials Network 1205 Study. Biol Blood Marrow Transplant. 2018 Oct;24(10):2145-2151. doi: 10.1016/j.bbmt.2018.04.014. Epub 2018 Apr 18. PMID 29679770
- [Background] Tulsky JA, Arnold RM, Alexander SC, Olsen MK, Jeffreys AS, Rodriguez KL, Skinner CS, Farrell D, Abernethy AP, Pollak KI. Enhancing communication between oncologists and patients with a computer-based training program: a randomized trial. Ann Intern Med. 2011 Nov 1;155(9):593-601. doi: 10.7326/0003-4819-155-9-201111010-00007. PMID 22041948
- [Background] Mitchell SL, Shaffer ML, Cohen S, Hanson LC, Habtemariam D, Volandes AE. An Advance Care Planning Video Decision Support Tool for Nursing Home Residents With Advanced Dementia: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2018 Jul 1;178(7):961-969. doi: 10.1001/jamainternmed.2018.1506. PMID 29868778
- [Background] Epstein AS, Volandes AE, Chen LY, Gary KA, Li Y, Agre P, Levin TT, Reidy DL, Meng RD, Segal NH, Yu KH, Abou-Alfa GK, Janjigian YY, Kelsen DP, O'Reilly EM. A randomized controlled trial of a cardiopulmonary resuscitation video in advance care planning for progressive pancreas and hepatobiliary cancer patients. J Palliat Med. 2013 Jun;16(6):623-31. doi: 10.1089/jpm.2012.0524. Epub 2013 Apr 22. PMID 23725233
- [Background] Reyna VF. A theory of medical decision making and health: fuzzy trace theory. Med Decis Making. 2008 Nov-Dec;28(6):850-65. doi: 10.1177/0272989X08327066. Epub 2008 Nov 17. PMID 19015287
- [Background] Derry HM, Maciejewski PK, Epstein AS, Shah MA, LeBlanc TW, Reyna V, Prigerson HG. Associations between Anxiety, Poor Prognosis, and Accurate Understanding of Scan Results among Advanced Cancer Patients. J Palliat Med. 2019 Aug;22(8):961-965. doi: 10.1089/jpm.2018.0624. Epub 2019 Feb 6. PMID 30724692
- [Background] Fenton JJ, Duberstein PR, Kravitz RL, Xing G, Tancredi DJ, Fiscella K, Mohile S, Epstein RM. Impact of Prognostic Discussions on the Patient-Physician Relationship: Prospective Cohort Study. J Clin Oncol. 2018 Jan 20;36(3):225-230. doi: 10.1200/JCO.2017.75.6288. Epub 2017 Nov 17. PMID 29148892
- [Background] de Meyrick J: The Delphi Method and Health Research. Health Education 103:7-16, 2003
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Background] Reyna VF, Nelson WL, Han PK, Pignone MP. Decision making and cancer. Am Psychol. 2015 Feb-Mar;70(2):105-18. doi: 10.1037/a0036834. PMID 25730718
- [Background] Singh S, Cortez D, Maynard D, Cleary JF, DuBenske L, Campbell TC. Characterizing the Nature of Scan Results Discussions: Insights Into Why Patients Misunderstand Their Prognosis. J Oncol Pract. 2017 Mar;13(3):e231-e239. doi: 10.1200/JOP.2016.014621. Epub 2017 Jan 17. PMID 28095172
- [Background] Shen MJ, Trevino KM, Prigerson HG. The interactive effect of advanced cancer patient and caregiver prognostic understanding on patients' completion of Do Not Resuscitate orders. Psychooncology. 2018 Jul;27(7):1765-1771. doi: 10.1002/pon.4723. Epub 2018 Apr 30. PMID 29611241
- [Background] Kurita K, Siegler EL, Reid MC, Maciejewski RC, Prigerson HG. It Is Not What You Think: Associations Between Perceived Cognitive and Physical Status and Prognostic Understanding in Patients With Advanced Cancer. J Pain Symptom Manage. 2018 Aug;56(2):259-263. doi: 10.1016/j.jpainsymman.2018.04.016. Epub 2018 May 10. PMID 29753102
- [Background] Cohen SM, Maciejewski RC, Shah MA, Trevino KM, Shen MJ, Maciejewski PK, Prigerson HG. Being present: oncologists' role in promoting advanced cancer patients' illness understanding. Cancer Med. 2018 Apr;7(4):1511-1518. doi: 10.1002/cam4.1389. Epub 2018 Feb 26. PMID 29479843
- [Background] Morse JM: Designing funded qualitative research. Handbook of qualitative research, Denzin and Lincoln (eds), Thousand Oaks, CA, Sage Publications, Inc:220-235, 1994
- [Background] Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975 Oct;23(10):433-41. doi: 10.1111/j.1532-5415.1975.tb00927.x. PMID 1159263
- [Background] van Vliet LM, Epstein AS. Current state of the art and science of patient-clinician communication in progressive disease: patients' need to know and need to feel known. J Clin Oncol. 2014 Nov 1;32(31):3474-8. doi: 10.1200/JCO.2014.56.0425. Epub 2014 Sep 29. No abstract available. PMID 25267758
- [Background] Gilligan T, Coyle N, Frankel RM, Berry DL, Bohlke K, Epstein RM, Finlay E, Jackson VA, Lathan CS, Loprinzi CL, Nguyen LH, Seigel C, Baile WF. Patient-Clinician Communication: American Society of Clinical Oncology Consensus Guideline. J Clin Oncol. 2017 Nov 1;35(31):3618-3632. doi: 10.1200/JCO.2017.75.2311. Epub 2017 Sep 11. PMID 28892432
- [Background] Back AL, Arnold RM. Discussing prognosis: "how much do you want to know?" talking to patients who are prepared for explicit information. J Clin Oncol. 2006 Sep 1;24(25):4209-13. doi: 10.1200/JCO.2006.06.007. No abstract available. PMID 16943539
- [Background] Hagerty RG, Butow PN, Ellis PM, Lobb EA, Pendlebury SC, Leighl N, MacLeod C, Tattersall MH. Communicating with realism and hope: incurable cancer patients' views on the disclosure of prognosis. J Clin Oncol. 2005 Feb 20;23(6):1278-88. doi: 10.1200/JCO.2005.11.138. PMID 15718326
- [Background] Jacobsen J, Brenner K, Greer JA, Jacobo M, Rosenberg L, Nipp RD, Jackson VA. When a Patient Is Reluctant To Talk About It: A Dual Framework To Focus on Living Well and Tolerate the Possibility of Dying. J Palliat Med. 2018 Mar;21(3):322-327. doi: 10.1089/jpm.2017.0109. Epub 2017 Oct 3. PMID 28972862
- [Background] McCambridge J, Witton J, Elbourne DR. Systematic review of the Hawthorne effect: new concepts are needed to study research participation effects. J Clin Epidemiol. 2014 Mar;67(3):267-77. doi: 10.1016/j.jclinepi.2013.08.015. Epub 2013 Nov 22. PMID 24275499
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of health care interventions: A theoretical framework and proposed research agenda. Br J Health Psychol. 2018 Sep;23(3):519-531. doi: 10.1111/bjhp.12295. Epub 2018 Feb 16. No abstract available. PMID 29453791
- [Background] Cohen SR, Mount BM, Strobel MG, Bui F. The McGill Quality of Life Questionnaire: a measure of quality of life appropriate for people with advanced disease. A preliminary study of validity and acceptability. Palliat Med. 1995 Jul;9(3):207-19. doi: 10.1177/026921639500900306. PMID 7582177
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Wright AA, Mack JW, Kritek PA, Balboni TA, Massaro AF, Matulonis UA, Block SD, Prigerson HG. Influence of patients' preferences and treatment site on cancer patients' end-of-life care. Cancer. 2010 Oct 1;116(19):4656-63. doi: 10.1002/cncr.25217. PMID 20572030
- [Background] Phillips RS, Wenger NS, Teno J, Oye RK, Youngner S, Califf R, Layde P, Desbiens N, Connors AF Jr, Lynn J. Choices of seriously ill patients about cardiopulmonary resuscitation: correlates and outcomes. SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. Am J Med. 1996 Feb;100(2):128-37. doi: 10.1016/s0002-9343(97)89450-8. PMID 8629646
- [Background] Mack JW, Block SD, Nilsson M, Wright A, Trice E, Friedlander R, Paulk E, Prigerson HG. Measuring therapeutic alliance between oncologists and patients with advanced cancer: the Human Connection Scale. Cancer. 2009 Jul 15;115(14):3302-11. doi: 10.1002/cncr.24360. PMID 19484795
- [Background] Davis TC, Long SW, Jackson RH, Mayeaux EJ, George RB, Murphy PW, Crouch MA. Rapid estimate of adult literacy in medicine: a shortened screening instrument. Fam Med. 1993 Jun;25(6):391-5. PMID 8349060
- [Background] Balboni TA, Prigerson HG, Balboni MJ, Enzinger AC, VanderWeele TJ, Maciejewski PK. A scale to assess religious beliefs in end-of-life medical care. Cancer. 2019 May 1;125(9):1527-1535. doi: 10.1002/cncr.31946. Epub 2019 Mar 2. PMID 30825390
- [Background] Canner PL. Covariate adjustment of treatment effects in clinical trials. Control Clin Trials. 1991 Jun;12(3):359-66. doi: 10.1016/0197-2456(91)90016-f. PMID 1651207
- [Background] Begg C, Cho M, Eastwood S, Horton R, Moher D, Olkin I, Pitkin R, Rennie D, Schulz KF, Simel D, Stroup DF. Improving the quality of reporting of randomized controlled trials. The CONSORT statement. JAMA. 1996 Aug 28;276(8):637-9. doi: 10.1001/jama.276.8.637. No abstract available. PMID 8773637
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] Schafer JL, Olsen MK. Multiple Imputation for Multivariate Missing-Data Problems: A Data Analyst's Perspective. Multivariate Behav Res. 1998 Oct 1;33(4):545-71. doi: 10.1207/s15327906mbr3304_5. PMID 26753828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out between 10/2020 and 6/2022 in outpatient GI and thoracic cancer clinics at Weill Cornell Medicine/New York Presbyterian. Patients were first chart-screened, and the treating oncologist's prognosis and permission were obtained for those potentially eligible. Patients were approached by phone (when COVID conditions required) or in clinic after an appointment with their oncologist.
Pre-assignment Details: Group assignment was not random, but was based on the arm of the participating patient's physician: GIST-trained or usual care. Screening for cognitive deficit and health literacy occurred prior to enrollment. Following enrollment, one patient withdrew due to time constraints and one was lost to follow-up.
Groups:
- Oncolo-GIST Arm - Patients: Patients assigned to this arm will will discuss scan results revealing progressive disease with an Oncolo-GIST trained physician.
  Oncolo-GIST: Behavioral: Oncolo-GIST Oncolo-GIST is a brief, manualized communication intervention that guides oncologists in "gist communication" by itemizing 4 key steps in the process of imparting prognostic information.
  Topic covered include:
  Principles of introducing prognosis in the setting of worsened scan results Coupling communicating realistic prognoses with psychological support (e.g., saying "average life-expectancy is months…" with emphasizing that the oncology team "will always provide care for you") Addressing informational needs and psychological reactions Applying proven techniques for supporting patients who are reluctant to discuss prognosis.
  The 4-step guide will include brief video-clips of demonstrating each "talking point" with a standardized patient, including ideal scenarios, common pitfalls to avoid, and how to respond to patient reactions that are particularly challenging, such as responding to optimism, death anxiety, and reliance on faith.
Period: Overall Study
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Started | 19 | 14 | 2 | 2
Completed Patient Baseline Assessment | 18 | 13 | 0 | 0
Had Progression on Scan | 13 | 12 | 0 | 0
Completed Post-scan Assessment | 13 | 11 | 0 | 0
Completed Physician Demographics Survey | 0 | 0 | 2 | 2
Completed Physician Oncolo-GIST Quiz | 0 | 0 | 2 | 0
Completed Physician Post-study Questionnaire | 0 | 0 | 2 | 2
Completed | 13 | 11 | 2 | 2
Not Completed | 6 | 3 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Did not have scan | 1 | 0 | 0 | 0
Not completed — In hospice care | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who completed the Baseline Survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians | Total
Number analyzed (Participants) | 18 | 13 | 2 | 2 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (12.6) | 61.5 (10.9) | 46.5 (7.8) | 55.5 (9.2) | 66.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 0 | 1 | 12
  Male | 10 | 10 | 2 | 1 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 3
  Not Hispanic or Latino | 17 | 11 | 2 | 2 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 0 | 4
  White | 14 | 11 | 0 | 2 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Cancer type (Diagnosis for patients; treatment specialty for physicians) [Count of Participants; unit: Participants]
  Gastrointestinal | 11 | 11 | 1 | 1 | 24
  Thoracic | 7 | 2 | 1 | 1 | 11
Religion [Count of Participants; unit: Participants]
  Christian | 12 | 7 | 0 | 0 | 19
  Jewish | 1 | 3 | 0 | 1 | 5
  Muslim | 1 | 1 | 0 | 0 | 2
  Other Religion | 0 | 2 | 1 | 0 | 3
  No Religion | 4 | 0 | 1 | 1 | 6
Education [Count of Participants; unit: Participants]
  Did Not Complete High School | 0 | 1 | 0 | 0 | 1
  High School | 5 | 0 | 0 | 0 | 5
  Some College | 3 | 2 | 0 | 0 | 5
  College Degree | 4 | 5 | 0 | 0 | 9
  Graduate Degree | 6 | 5 | 2 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Prognostic Understanding
Description: Changes in illness understanding by patients as measured by three items from the investigator's validated 4-item assessment will be compared between groups at baseline and post-scan follow-up. The assessment asks three questions that assess patients' recognition of their incurable disease status, knowledge of the advanced stage of their disease, and expectation to live months as opposed to years. Responses are coded 1 or 0 to indicate the presence or absence of each of these element. These four indicators are then added together to construct summary scores (possible range, 0 to 3). Differences between pre- and post-scan visit illness understanding scores (possible range, -3 to 3) are used to define changes in illness understanding by a patient between the pre- and post-scan visit interviews. Higher total scores represent an increase in prognostic understanding. Lower scores represent a decrease in understanding.
Time Frame: Baseline; week after scan. 2- and - 4-month assessments were ultimately not done as participants preferred not to commit to follow-up.
Population: 1 patient on the Oncolo-GIST arm was not analyzed due to not having completed the post-scan visit interview. Not relevant to Physician arm participants. The investigators did not include one item from the validated 4-item scale (terminal illness acknowledgement) in the follow-up assessment due to technical error, and so the measure was limited to the three items for which there was follow-up data. 2- and - 4-month assessments were not done as participants preferred not to commit to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Oncolo-GIST Arm - Patients: Patients assigned to this arm will will discuss scan results revealing progressive disease with an Oncolo-GIST trained physician.
  Oncolo-GIST: Behavioral: Oncolo-GIST Oncolo-GIST is a brief, manualized communication intervention that guides oncologists in "gist communication" by itemizing 4 key steps in the process of imparting prognostic information.
  Topics covered include:
  Principles of introducing prognosis in the setting of worsened scan results Coupling communicating realistic prognoses with psychological support (e.g., saying "average life-expectancy is months…" with emphasizing that the oncology team "will always provide care for you") Addressing informational needs and psychological reactions Applying proven techniques for supporting patients who are reluctant to discuss prognosis.
  The 4-step guide will include brief video-clips of demonstrating each "talking point" with a standardized patient, including ideal scenarios, common pitfalls to avoid, and how to respond to patient reactions that are particularly challenging, such as responding to optimism, death anxiety, and reliance on faith.
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Number analyzed (Participants) | 12 | 11 | 0 | 0
units on a scale | 0.58 (1.00) | 0.18 (1.25) |  |

2. Secondary Outcome: Patient Quality of Life
Description: Quality of life of patients, as measured by the McGill Quality of Life Questionnaire, will be compared between groups at one-week, two-month and 4-month follow up assessments (T2, T3, and T4). This questionnaire contains 16 items and each item uses a 10-point scale, where 0 is desirable and 10 is undesirable. Separate sub-scales scoring for global, physical, psychological, emotional and existential well-being, are determined by taking the mean of the associated items. The score for overall quality of life is determined by taking the mean of all the sub-scales. Higher total scores represent better quality of life. Lower scores represent worse better quality of life.
Time Frame: Day 1, within one week, 2 months, 4 month
Population: Data was not collected for this measure.
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Whether or Not a Do Not Resuscitate Was Ordered by Patient
Description: Whether or not a Do Not Resuscitate (DNR) was ordered by the patient, as determined by a medical chart abstraction, will be compared between groups at 2-month and 4-month follow up assessments (T4). This will be scored as either a 0, if there was no DNR ordered, or a 1 if there was a DNR ordered.
Time Frame: 1 week post-scan, 2 months post-scan, 4 months post-scan.
Population: All patients who completed follow-up assessments and therefore had a medical chart review. This measure is not relevant to physician participants. 4-month assessments were ultimately not done, as participants preferred not to commit to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Number analyzed (Participants) | 13 | 11 | 0 | 0
Participants
  1 Week Post-Scan | 0 | 0 | 0 | 0
  2 months Post-Scan | 0 | 0 |  |

4. Secondary Outcome: Treatment and Care Received
Description: Methods of treatment and care received by patients, as determined from a medical chart abstraction, will be compared between groups at 2-month and 4-month follow up assessments (T4). Types of care include palliative care, hospice and hospitalization. Types of treatment include chemotherapy drugs, narcotic pain medication and radiation therapy.
Time Frame: 1 week post-scan, 2 months post-scan, 4 months post-scan.
Population: Data collection for this outcome was discontinued when the assessment at 4 months was eliminated. No data was collected at 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Number analyzed (Participants) | 10 | 7 | 0 | 0
Participants
  1 Week Post-Scan : Patients enrolled in hospice care | 0 | 0 |  |
  1 Week Post-Scan : Patients who had had a palliative care consult | 0 | 0 |  |
  1 Week Post-Scan: Patients who had been hospitalized within the past week. | 0 | 1 |  |
  1 Week Post-Scan: Patients who were receiving chemotherapy | 10 | 6 |  |
  1 Week Post-Scan: Patients who were receiving radiation therapy | 1 | 1 |  |
  1 Week Post-Scan: Patients who were receiving narcotic pain medication | 7 | 5 |  |
  2 Months Post-Scan : Patients enrolled in hospice care | 0 | 0 |  |
  2 Months Post-Scan : Patients who had had a palliative care consult | 1 | 0 |  |
  2 Months Post-Scan: Patients who had been hospitalized within the past week. | 0 | 0 |  |
  2 Months Post-Scan: Patients who were receiving chemotherapy | 10 | 7 |  |
  2 Months Post-Scan: Patients who were receiving radiation therapy | 0 | 0 |  |
  2 Months Post-Scan: Patients who were receiving narcotic pain medication | 7 | 5 |  |

5. Secondary Outcome: Patient Performance Status
Description: as for outcome 4
Time Frame: 1 week post-scan, 2 months post-scan.
Population: Data was not collected for this measure. Patient performance status was not noted in the majority of patients' charts, and where it was noted, physicians used differing scales.
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Post Hoc Outcome: Change in Physician-Patient Therapeutic Alliance as Measured by the Human Connection Scale
Description: Changes in 11-item Human Connection Scale (Mack et al., 2009) total score and individual item scores after scan discussion. Total scores have a range of 0-44 and are calculated by summing individual item scores from the 11 items on the assessment. Individual items are scored from 0-4. In both cases, higher scores mean a better outcome: a stronger physician-patient therapeutic alliance. Change scores are calculated by subtracting the mean at the week after scan (T1) from the mean at baseline. A positive change indicates a better outcome (strengthening of the therapeutic alliance), whereas a negative change indicates a worse outcome (weakening of the therapeutic alliance).
Time Frame: Baseline, week after scan.
Population: All participants who completed follow-up assessments. This measure is not relevant to physician participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Number analyzed (Participants) | 13 | 11 | 0 | 0
score on a scale
  Change in Human Connection Scale total score | -1.00 (1.63) | 0.14 (1.57) |  |
  Change in individual item: Likes oncologist | 0.00 (0.00) | 0.00 (0.00) |  |
  Change in individual item: trusts oncologist | 0.00 (0.00) | 0.00 (0.00) |  |
  Change in individual item: Oncologist is concerned about your quality of life. | 0.23 (0.44) | 0.27 (1.01) |  |
  Change in individual item: doctor asks how you are coping with cancer. | 0.15 (0.80) | 0.09 (1.14) |  |
  Change in individual item: Doctor asks how family members are coping with illness. | 0.50 (1.27) | 0.20 (0.63) |  |
  Change in individual item: Feels comfortable asking doctor questions. | -0.42 (0.90) | 0.00 (0.00) |  |
  Change in individual item: Oncologist takes the time to listen to concerns. | -0.08 (0.64) | 0.00 (0.45) |  |
  Change in individual item: Oncologist sees you as a whole person. | -0.08 (0.28) | 0.00 (0.00) |  |
  Change in individual item: Oncologist cares about you. | -0.08 (0.49) | 0.00 (0.00) |  |
  Change in individual item: Oncologist is honest with you. | 0.00 (0.47) | 0.00 (0.00) |  |
  Change in individual item: Oncologist offers hope. | -0.22 (0.67) | 0.11 (0.33) |  |

7. Post Hoc Outcome: Change in Anxiety and Depression as Measured by the Hospital Anxiety and Depression Scale Anxiety and Depression Subscores
Description: Changes in Hospital Anxiety and Depression Scale Anxiety and Depression subscores, each with a minimum of 0 and maximum of 21, with a higher score meaning a worse outcome and a negative change between timepoints indicating improvement.
Time Frame: Baseline, week after scan
Population: All patients who completed follow-up assessments. This measure is not relevant to physician participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
Number analyzed (Participants) | 13 | 11 | 0 | 0
score on a scale
  Anxiety subscore change | 0.64 (2.50) | 0.40 (1.43) |  |
  Depression subscore change | 1.64 (3.80) | 2.45 (3.14) |  |

ADVERSE EVENTS:
Time Frame: 2 years, 1 month
Description: For the purpose of this study, an AE is defined as a participant experiencing severe psychological distress, regardless of attribution. Serious Adverse Events (SAEs) were not monitored or assessed. All-Cause Mortality and Other [Not Including Serious] Adverse Events were not monitored/assessed for physician participants.
Arm/Group | Oncolo-GIST Arm - Patients | Usual Care Arm - Patients | Oncolo-GIST Arm - Physicians | Usual Care Arm - Physicians
All-Cause Mortality (participants affected / at risk) | 1/19 | 1/14 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/19 | 0/14 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Enrollment was lower than planned, limiting statistical power and generalizability of the results. Due to technical error, some measures, including the McGill Quality of Life scale and a question about terminal illness understanding from the patient assessments, were omitted. We also modified the protocol to eliminate two planned follow-ups to increase acceptability. Therefore, we did not analyze most planned secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT04179305/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT04179305/ICF_002.pdf